CLINICAL TRIAL: NCT00005908
Title: A Pilot Trial of Sequential Primary (Neoadjuvant) Combination Chemotherapy With Docetaxel/Capecitabine (TX) and Doxorubicin/Cyclophosphamide (AC) in Primary Breast Cancer With Evaluation of Chemotherapy Effects on Gene Expression
Brief Title: Primary Chemotherapy With Docetaxel-Capecitabine and Doxorubicin-Cyclophosphamide in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jo Anne Zujewski, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000149; 00-C-0149; NCT00020241 (obsolete NCT alias)
Record Dates: First submitted 2000-06-13; First posted 2000-06-14 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: cDNA Microarray; Stage II and Stage III Breast Cancer; Biological Response; Molecular Profiling; Fine Needle Aspirate; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine; Anastrozole; Cyclophosphamide; Doxorubicin; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose A-Cohort 1-Arm 1-Docetaxel & Capecitabine (Experimental): Docetaxel 75 mg/m^2 intravenous day 1, capecitabine 1000 mg/m^2 orally twice daily day 2-15 for 4 cycles
  Interventions: Drug: Docetaxel - Dose A; Drug: Anastrozole; Drug: cyclophosphamide; Drug: Doxorubicin hydrochloride; Drug: Tamoxifen Citrate; Drug: Capecitabine - Dose A
- Dose B-Cohort 2-Arm 2 Reduced dose-Docetaxel & Capecitabine (Experimental): Docetaxel 60 mg/m^2 intravenous day 1, capecitabine 937.5 mg/m^2 orally twice daily day 2-15 for 4 cycles
  Interventions: Drug: Anastrozole; Drug: cyclophosphamide; Drug: Docetaxel - Dose B; Drug: Doxorubicin hydrochloride; Drug: Tamoxifen Citrate; Drug: Capecitabine - Dose B

INTERVENTIONS:
Drug: Docetaxel - Dose A — Dose A-Cohort 1 Docetaxel 75 mg/m^2 intravenous day 1
  Other Names: Taxotere/Xeloda
  Arms: Dose A-Cohort 1-Arm 1-Docetaxel & Capecitabine
Drug: Anastrozole — 1 mg orally daily for five years
  Other Names: Arimidex
Drug: cyclophosphamide — 600 mg/m^2 will be diluted in 100 mL 0.9% normal saline (NS) and administered intravenously over 30 minutes on day 1
  Other Names: Cytoxan
Drug: Docetaxel - Dose B — Dose B - Cohort 2 Docetaxel 60 mg/m^2 intravenous day 1
  Other Names: Taxotere
  Arms: Dose B-Cohort 2-Arm 2 Reduced dose-Docetaxel & Capecitabine
Drug: Doxorubicin hydrochloride — 60 mg/m^2 will be administered as a slow intravenous push on day 1
  Other Names: Adriamycin
Drug: Tamoxifen Citrate — 20 mg/day orally for five years
  Other Names: Nolvadex
Drug: Capecitabine - Dose B — Dose B - Cohort 2 capecitabine 937.5 mg/m^2 orally twice daily day 2-15
  Arms: Dose B-Cohort 2-Arm 2 Reduced dose-Docetaxel & Capecitabine
Drug: Capecitabine - Dose A — capecitabine 1000 mg/m^2 orally twice daily day 2-15 for 4 cycles
  Arms: Dose A-Cohort 1-Arm 1-Docetaxel & Capecitabine

SUMMARY:
This study will assess the usefulness of a technique called complementary deoxyribonucleic acid (cDNA) microarray-an examination of a wide array of genes to identify disease-associated patterns-for measuring tumor response to chemotherapy in breast cancer patients. The study will look for "markers" that can help select the most effective type of chemotherapy. It will also evaluate the safety and effectiveness of a new drug combination of capecitabine and docetaxel.

Patients age 18 years and older with stage II or III breast cancer whose tumor is 2 centimeters or larger may be eligible for this study. Those enrolled will be treated with surgery, standard chemotherapy using doxorubicin (Adriamycin) and cyclophosphamide (Cytoxan), and the capecitabine and docetaxel combination.

Patients will have a physical examination, mammogram and magnetic resonance imaging to evaluate their tumor before beginning treatment. They will then have four 21-day treatment cycles of docetaxel and capecitabine, as follows: docetaxel intravenously (through a vein) on day 1 and capecitabine pills (by mouth) twice a day from days 2 through 15. No drugs will be given from days 16 through 21. This regimen will be repeated four times, after which the tumor will be re-evaluated by physical examination, mammogram, and magnetic resonance imaging.

Patients will then have surgery to remove the cancer-either lumpectomy with removal of the underarm lymph nodes; mastectomy and removal of the underarm lymph nodes; or modified radical mastectomy. After recovery, they will have four more cycles of chemotherapy, this time with a doxorubicin and cyclophosphamide. Both drugs will be given intravenously on day 1 of four 21-day cycles.

Some patients who had a mastectomy (depending on their tumor characteristics and whether tumor cells were found in their lymph nodes) and all those who had a lumpectomy will also have radiation therapy. Patients with hormone receptor-positive tumors will also receive tamoxifen treatment for 5 years.

In addition to the above procedures, all patients will have tumor biopsies (removal of a small piece of tumor tissue) before beginning treatment, on day 1 of cycle 1, before cycle 2, and at the time of surgery, and physical examinations, chest X-rays, bone scans, computerized tomography (CT) scans, electrocardiograms, multi-gated acquisition scan-MUGA (nuclear medicine test of cardiac function) or echocardiograms of heart function, mammograms and blood tests at various times during the study. Patients will be followed at National Institutes of Health (NIH) for 3 years after diagnosis with physical examinations, blood tests, X-rays, and computed tomography (CT) scans.

Although it is not known whether this treatment will help an individual patient's cancer, possible benefits are tumor shrinkage and decreased risk of disease recurrence. In addition, the information gained about genetic changes after chemotherapy will help determine if additional studies on the use of cDNA microarray to measure tumor response are warranted.

DETAILED DESCRIPTION:
This phase II trial in patients with stage II and stage III breast cancer will test the feasibility of using cDNA microarray as a measure of a tumor's biological response to chemotherapeutic agents by characterizing the cDNA expression patterns in breast cancer before and after primary chemotherapy. Thirty-six patients receive docetaxel/capecitabine induction chemotherapy followed by surgery and doxorubicin/cyclophosphamide adjuvant therapy (TX/AC). We will determine the response rate of TX induction therapy and the toxicities of the sequential combinations (TX/AC). We will also obtain tumor tissue for correlative biological determinations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Stage II or III breast cancer with a tumor size of greater than 2 cm. Patients with a previous biopsy are eligible provided adequate tumor tissue remains for biopsy in this study.

At least 18 years of age.

Adequate hematopoietic function as defined by absolute neutrophil count greater than 1200/mm^3 and platelet count greater than 100,000/mm^3.

Adequate renal function as defined by creatinine less than 1.6 mg/dL.

Adequate hepatic function as defined by total (T.) bilirubin less than 1.4 mg/dL and serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvic transaminase (SGPT) less than 1.5 times the upper limit of normal and alkaline phosphatase less than 2.5 times upper limit of normal

Zubrod Performance status 0-2.

EXCLUSION CRITERIA:

Medical or psychiatric condition that, in the opinion of the Principal Investigator, would preclude chemotherapy administration. Patients may be evaluated by psychiatry or medical subspecialties as appropriate.

Pregnant or lactating women

Known bleeding disorders

Hypersensitivity to Tween 80 (Polysorbate)

Cardiac ejection fraction below normal limits, myocardial infarction within the past 12 months, or symptomatic arrhythmia requiring medical intervention.

Prior chemotherapy or hormonal therapy for breast cancer. Patients treated with hormonal chemoprevention (tamoxifen or raloxifene) will be eligible.

Active malignancy diagnosed within the last 5 years. (Cervical cancer or non-melanomatous skin cancer that has been treated with curative intent will be eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnne Zujewski, M.D., Principal Investigator — National Cancer Institute (NCI), National Institutes of Health (NIH)
Locations (1):
- National Naval Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Elledge RM, Gray R, Mansour E, Yu Y, Clark GM, Ravdin P, Osborne CK, Gilchrist K, Davidson NE, Robert N, et al. Accumulation of p53 protein as a possible predictor of response to adjuvant combination chemotherapy with cyclophosphamide, methotrexate, fluorouracil, and prednisone for breast cancer. J Natl Cancer Inst. 1995 Aug 16;87(16):1254-6. doi: 10.1093/jnci/87.16.1254. No abstract available. PMID 7563172
- [Background] MacGrogan G, Mauriac L, Durand M, Bonichon F, Trojani M, de Mascarel I, Coindre JM. Primary chemotherapy in breast invasive carcinoma: predictive value of the immunohistochemical detection of hormonal receptors, p53, c-erbB-2, MiB1, pS2 and GST pi. Br J Cancer. 1996 Nov;74(9):1458-65. doi: 10.1038/bjc.1996.565. PMID 8912545
- [Background] Harvey JM, Clark GM, Osborne CK, Allred DC. Estrogen receptor status by immunohistochemistry is superior to the ligand-binding assay for predicting response to adjuvant endocrine therapy in breast cancer. J Clin Oncol. 1999 May;17(5):1474-81. doi: 10.1200/JCO.1999.17.5.1474. PMID 10334533
- [Result] Lebowitz PF, Eng-Wong J, Swain SM, Berman A, Merino MJ, Chow CK, Venzon D, Zia F, Danforth D, Liu E, Zujewski J. A phase II trial of neoadjuvant docetaxel and capecitabine for locally advanced breast cancer. Clin Cancer Res. 2004 Oct 15;10(20):6764-9. doi: 10.1158/1078-0432.CCR-04-0976. PMID 15501952
- [Result] Korde LA, Lusa L, McShane L, Lebowitz PF, Lukes L, Camphausen K, Parker JS, Swain SM, Hunter K, Zujewski JA. Gene expression pathway analysis to predict response to neoadjuvant docetaxel and capecitabine for breast cancer. Breast Cancer Res Treat. 2010 Feb;119(3):685-99. doi: 10.1007/s10549-009-0651-3. PMID 20012355
- See also: RECIST — http://ctep.cancer.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose A-Cohort 1-Arm 1-Docetaxel & Capecitabine: Docetaxel 75 mg/m^2 intravenous day 1, capecitabine 1000 mg/m^2 orally twice daily day 2-15 for 4 cycles Once the dose was deemed to be too toxic, subsequent patients were enrolled on dose B.
- Dose B-Cohort 2-Arm 2 Reduced Dose-Docetaxel & Capecitabine: Docetaxel 60 mg/m^2 intravenous day 1 capecitabine 937.5 mg/m^2 orally twice daily day 2-15
Period: Overall Study
Arm/Group | Dose A-Cohort 1-Arm 1-Docetaxel & Capecitabine | Dose B-Cohort 2-Arm 2 Reduced Dose-Docetaxel & Capecitabine
Started | 10 | 20
Completed | 9 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel/Capecitabine - A & B: Docetaxel/Capecitabine - A- Docetaxel 75 mg/m^2 intravenous day 1,capecitabine 1000 mg/m^2 orally twice daily day 2-15 for 4 cycles. Docetaxel/Capecitabine - B- Docetaxel 60 mg/m^2 intravenous day 1 capecitabine 937.5 mg/m^2 orally twice daily day 2-15
Arm/Group | Docetaxel/Capecitabine - A & B
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 15
  African American | 6
  Asian | 6
  Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 6 years
Measure: Number; unit: Participants
Arm/Group | Dose A-Cohort 1-Arm 1-Docetaxel & Capecitabine | Dose B-Cohort 2-Arm 2 Reduced Dose-Docetaxel & Capecitabine
Number analyzed (Participants) | 9 | 20
Participants | 9 | 20

2. Primary Outcome: Overall Clinical Response Rate
Description: Overall response rate is defined as the percentage of participants with a CR (complete disappearance of all target lesions), PR (a 30% decrease in the sum of the longest diameter of target lesions) determined by clinical measurements per the Response Evaluation Criteria in Solid Tumors (RECIST) and/or a complete pathologic response (disappearance of all invasive tumor pathologically or presence of ductal carcinoma in situ) per the Chevallier criteria. For details about the RECIST or Chevallier criteria see the protocol link module.
Time Frame: 6 years
Population: Combined data from 2 dose levels in 29 evaluable patients.
Measure: Number; unit: Percentage of participants
Groups:
- Dose A & B-Cohort 1 & 2-Arm 1& 2-Docetaxel & Capecitabine: Docetaxel 75 mg/m^2 intravenous day 1, capecitabine 1000 mg/m^2 orally twice daily day 2-15 for 4 cycles Docetaxel 60 mg/m^2 intravenous day 1 capecitabine 937.5 mg/m^2 orally twice daily day 2-15
Arm/Group | Dose A & B-Cohort 1 & 2-Arm 1& 2-Docetaxel & Capecitabine
Number analyzed (Participants) | 29
Percentage of participants
  Complete Response | 31
  Partial Response | 59
  Complete pathologic response | 10

3. Primary Outcome: Complementary Deoxyribonucleic Acid (cDNA) Expression
Description: Patients were classified as responders or non-responders based on change in tumor size by clinical exam and pathologic response.For instance, patients with a pathological complete response, micro-invasive disease at surgery, or clinical complete response after four cycles of treatment were considered responders. Changes in gene expression associated with treatment was assessed before/after chemotherapy. All gene expression summary intensities below 50 were thresholded to the value of 50 and genes showing variability significantly smaller than the median gene variability were screened out.
Time Frame: 6 years
Measure: Number; unit: Participants
Groups:
- Dose B-Cohort 2-Arm 2 Reduced Dose-Docetaxel & Capecitabine: Docetaxel 60 mg/m^2 intravenous day 1, capecitabine 937.5 mg/m^2 orally twice daily day 2-15
Arm/Group | Dose A-Cohort 1-Arm 1-Docetaxel & Capecitabine | Dose B-Cohort 2-Arm 2 Reduced Dose-Docetaxel & Capecitabine
Number analyzed (Participants) | 10 | 20
Participants
  Responders | 8 | 7
  Non-responders | 2 | 13

4. Primary Outcome: Number of Participants, e.g. Responders and Non-responders With a Percent Change in Expression Patterns After Chemotherapy With Changes in Expression Patterns After Chemotherapy in Preclinical Models
Description: as for outcome 3
Time Frame: 6 years
Population: Specimens from 21 patients. Analysis was "per protocol" and included only those patients with adequate RNA (ribonucleic acid) for analysis. Since both had the same intervention, the sample size was small, and a dose response was not expected, all patients were analyzed together.
Measure: Number; unit: Participants
Groups:
- Dose A & B-Cohort 1 & 2-Arm 1 & 2-Docetaxel & Capecitabine: Docetaxel 75 mg/m^2 intravenous day 1, capecitabine 1000 mg/m^2 orally twice daily day 2-15 for 4 cycles
Arm/Group | Dose A & B-Cohort 1 & 2-Arm 1 & 2-Docetaxel & Capecitabine
Number analyzed (Participants) | 21
Participants
  Responders | 8
  Non-responders | 13

ADVERSE EVENTS:
Time Frame: 6 years
Description: CTC version 2.0 criteria for adverse event report. If a specific description was not available in the standard 'CTC" criteria the event was categorized by the major class and "other".
Groups:
- Docetaxel/Capecitabine - A & B: Docetaxel/Capecitabine - A- Docetaxel 75 mg/m^2 intravenous day 1,capecitabine 1000 mg/m^2 orally twice daily day 2-15 for 4 cycles. Docetaxel/Capecitabine - B- Docetaxel 60 mg/m2 intravenous day 1 capecitabine 937.5 mg/m2 orally twice daily day 2-15
Arm/Group | Docetaxel/Capecitabine - A & B
Serious Adverse Events (participants affected / at risk) | 29/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel/Capecitabine - A & B (N=30)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 5 (5)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 3 (3)
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 2 (2)
Hand/foot skin reaction (Skin and subcutaneous tissue disorders) | 13 (16)
Neuropathy-sensory (Nervous system disorders) | 1 (1)
Infection, Other (Infections and infestations) | 5 (5)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) — (fever of unknown origin without clinically or microbiologically documented infection)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (13)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 4 (4)
Infection without neutropenia (Infections and infestations) | 2 (3)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1)
Leukocytes (total WBC) (Investigations) | 12 (44)
Lymphatics (Blood and lymphatic system disorders) | 1 (1)
Mood alteration-depression (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 26 (135)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SGOT (AST) (Investigations) | 1 (1)
SGPT (ALT) (Investigations) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal/mucositis) (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound-infectious (Injury, poisoning and procedural complications) | 1 (1)
Wound-non-infectious (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel/Capecitabine - A & B (N=30)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 10 (24)
Memory loss (Nervous system disorders) | 3 (3)
Abdominal pain or cramping (Gastrointestinal disorders) | 4 (6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 (5)
Allergy-Other (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (26)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 7 (11)
Bilirubin (Investigations) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (9)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 7 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine (Investigations) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dermatitis, focal (associated with high-dose chemotherapy and bone marrow transplant) (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2)
Dyspepsia/heartburn (Gastrointestinal disorders) | 2 (2)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (General disorders) | 2 (2)
Fatigue (lathargy, malaise, asthenia) (General disorders) | 18 (53)
Fever (in absence of neutropenia, where neutropenia is defined as AGC<1.0x109/L) (General disorders) | 2 (4)
Flatulence (Gastrointestinal disorders) | 2 (3)
GI-Other (Gastrointestinal disorders) | 2 (2)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 11 (26)
Headache (Psychiatric disorders) | 8 (9)
Hearing-Other (Ear and labyrinth disorders) | 1 (1)
Hematologic-Other (Blood and lymphatic system disorders) | 2 (2)
Hematuria (in absence of vaginal bleeding) (Renal and urinary disorders) | 1 (2)
Hemoglobin (hgb) (Investigations) | 9 (39)
Hot flashes/flashes (Vascular disorders) | 16 (22)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (36)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (13)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 11 (18)
Infection, Other (Infections and infestations) | 3 (3)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 3 (3)
Leukocytes (total WBC) (Investigations) | 21 (103)
Libido (Reproductive system and breast disorders) | 4 (4)
Lymphatics (Blood and lymphatic system disorders) | 4 (4)
Lymphatics-Other (Blood and lymphatic system disorders) | 1 (1)
Metabolic-Other (Metabolism and nutrition disorders) | 1 (1)
Mood alteration-anxiety/agitation (Psychiatric disorders) | 7 (9)
Mood alteration-depression (Psychiatric disorders) | 8 (12)
Mouth dryness (Gastrointestinal disorders) | 2 (2)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 9 (17)
Nail changes (Skin and subcutaneous tissue disorders) | 10 (11)
Nausea (Gastrointestinal disorders) | 12 (34)
Neuropathy motor (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 25 (71)
Ocular-Other (Eye disorders) | 1 (1)
Pain-Other (General disorders) | 9 (13)
Palpitation (Cardiac disorders) | 2 (3)
Phlebitis (superficial) (Vascular disorders) | 2 (2)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 3 (3)
Platelets (Investigations) | 3 (5)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Renal/GU-Other (Renal and urinary disorders) | 1 (2)
Sexual/reproductive function-Other (Reproductive system and breast disorders) | 5 (5)
SGOT (AST) (Metabolism and nutrition disorders) | 5 (9)
SGPT (ALT) (Metabolism and nutrition disorders) | 6 (12)
Skin-Other (Skin and subcutaneous tissue disorders) | 3 (3)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 13 (22)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT (Gastrointestinal disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Syndromes-Other (General disorders) | 1 (1)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 10 (21)
Tearing (watery eyes) (Eye disorders) | 9 (12)
Vaginal bleeding (Blood and lymphatic system disorders) | 1 (3)
Vision-blurred vision (Eye disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 8 (21)
Weight loss (Investigations) | 1 (1)
Neuro-sensory (Nervous system disorders) | 10 (17)
Anorexia (Gastrointestinal disorders) | 8 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No